CLINICAL TRIAL: NCT02171169
Title: Retrospective, Multicenter Clinical Evaluation of Health Economic Drivers and Complications for Two Lumbar Fusion Procedures
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Baxano Surgical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-07875
Record Dates: First submitted 2014-06-19; First posted 2014-06-24 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Spinal Stenosis; Spondylolisthesis; Degenerative Disc Disease (DDD)
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Transsacral lumbar interbody fusion
- Transforaminal lumbar interbody fusion

SUMMARY:
The purpose of this retrospective data review is to evaluate the health economic drivers and complications of two surgical procedures: transsacral lumbar interbody fusion and transforaminal lumbar interbody fusion when used in conjunction with bilateral supplemental screw fixation as an adjunct to fusion. Devices used in both systems are cleared for use and comply with US regulations and requirements.

DETAILED DESCRIPTION:
Study Objective:

The study objective is to demonstrate via retrospective data review the relative value of two lumbar fusion procedures: transsacral lumbar interbody fusion and the transforaminal lumbar interbody fusion when used in conjunction with bilateral supplemental screw fixation as an adjunct to fusion. Subject candidates are those who had required fusion at L5-S1 where this was the only lumbar level treated for spinal stenosis, spondylolisthesis, or degenerative disc disease (DDD).

Consecutive subjects who were treated with the transsacral lumbar interbody fusion or transforaminal lumbar interbody fusion procedure at least 1 year (- 2 months) prior to the date the data is collected will be evaluated.

Study Design, Endpoints:

Primary Endpoint:

Safety: Incidence of reported adverse events, including those requiring medical intervention, by 3 months post-operative.

Secondary Endpoints:

Health Economic: Operative measures, including the direct and surrogate measurement of estimated blood loss, anesthesia time, transfusions, length of surgery and time to hospital discharge, as applicable.

Health Economic: Comparative hospital data (from time of admission through time of discharge)

Clinical Effectiveness: A decrease in back pain compared to baseline at 3 months (+/-2 weeks) as measured by Visual Analog Scale (VAS).

Clinical Effectiveness: A decrease in disability compared to baseline at 3 months (+/-2 weeks) as measured by the Oswestry Disability Index (ODI).

Study Design, Enrollment:

Approximately 200 subjects will be enrolled in this study, 100 subjects who have been treated with transsacral lumbar interbody fusion and 100 subjects who have been treated with transforaminal lumbar interbody fusion.

Study Design, Analyses:

The retrospective clinical evaluation will collect and compare results for the procedure transsacral lumbar interbody fusion versus transforaminal lumbar interbody fusion as defined by the primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 years or older
* Male or Female subject that had previously received transsacral single-level procedure when used in conjunction with bilateral pedicle screw fixation or TLIF single-level procedure with bilateral supplemental screw fixation (e.g. pedicle screws, anterior devices with screw anchoring, anterior lumber plates) as an adjunct to fusion at L5-S1 to treat spinal stenosis, spondylolithesis or degenerative disc disease (DDD)
* Subject that was treated no less than 1 year (-2 months) prior to this evaluation with a transsacral or TLIF procedure by participating surgeons

Exclusion Criteria:

* Subject had history of previous back operations at the time of the index procedure
* Subject had extraspinal cause of back pain or sciatica at the time of the index procedure
* Severe scoliosis in the lumbar region
* Subject was or is currently involved in active litigation
* Subject that had a diagnosis and received a transsacral or TLIF procedure at L5-S1 levels and did not require treatment at any other lumbar levels at the time of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject candidates are those that have been treated with either the transsacral or transforaminal lumbar interbody fusion procedure at least one year prior to this evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Safety | 3 months post-operative
  Incidence of reported adverse events, including those requiring medical intervention.

SECONDARY OUTCOMES:
Health Economic | Up to 3 months post-operative
  Operative measures including the direct and surrogate measurement of estimated blood loss, anesthesia time, transfusions, length of surgery and time to hospital discharge.
  Comparative hospital data
Clinical Effectiveness | 3 months post-operative
  A decrease in back pain compared to baseline at 3 months as measured by Visual Analog Scale A decrease in disability compared to baseline at 3 months as measure by the Oswestry Disability Index

CONTACTS AND LOCATIONS:
Overall Officials: Peter Whang, MD, Study Director — Yale University
Locations (3):
- United States (3):
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Michigan Spine Institute, Waterford, Michigan
  - University Hospitals Case Medical Center, Cleveland, Ohio